CLINICAL TRIAL: NCT04015973
Title: A Randomised Controlled Trial of a Pre-operative High Energy Diet for the Prevention of Organ Injury in Cardiac Surgery: The PRE-OP ENERGY Trial
Brief Title: The PRE-OP ENERGY Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0668; 246009 (Registry Identifier: IRAS); 18/EM/0254 (Other: REC East Midlands - Leics Central)
Record Dates: First submitted 2019-05-20; First posted 2019-07-11 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Valve Disease; Coronary Artery Disease; Organ Failure, Multiple
MeSH Terms: conditions — Heart Valve Diseases; Coronary Artery Disease; Multiple Organ Failure

STUDY DESIGN:
Intervention Model Description: Unblinded randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Control (No Intervention): Standard Care
- Group B: High energy diet (Experimental): High energy diet for 8-12 weeks pre-surgery
  Interventions: Dietary Supplement: High energy diet

INTERVENTIONS:
Dietary Supplement: High energy diet — An overfeeding regime of 135% required energy intake per day, set from baseline energy requirements consisting of high (saturated) fat snacks, added to the usual diet, supervised by a dietitian.
  Arms: Group B: High energy diet

SUMMARY:
The PRE-OP ENERGY Trial proposes to test the overarching hypothesis that a pre-surgery high energy diet will protect patients against organ damage during cardiac surgery with cardiopulmonary bypass.

DETAILED DESCRIPTION:
PRE-OP ENERGY is a single centre, unblinded, parallel group, randomised controlled trial of a pre-operative high energy diet, versus a control group receiving standard care.

The trial will test a number of specific hypotheses:

1. A pre-surgery high energy diet will protect against post-cardiac surgery organ failure by altering the pre-surgery cardiometabolic state, a process referred to as 'metabolic preconditioning'.
2. The effects of the trial intervention will not be attributable to changes in frailty, activity or baseline organ dysfunction.
3. The trial intervention will not result in long-term adverse changes in cardiometabolic status.
4. Metabolic preconditioning will confer protection against post-cardiac surgery kidney injury by increasing the expression of genes that promote renal tubular homeostasis.
5. Metabolic preconditioning will confer protection against post-cardiac surgery myocardial injury by increasing the expression of genes that promote myocardial mitochondrial homeostasis via effects on chromatin histone deacetylation.
6. Metabolic preconditioning will confer protection against post-cardiac surgery endothelial dysfunction by increasing the expression of genes that promote endothelial homeostasis.

ELIGIBILITY:
Inclusion Criteria:

ALL of the following:

* Adult cardiac surgery patients (≥18 years) undergoing cardiac surgery (CABG, Valve, or CABG and Valve) with cardiopulmonary bypass.
* BMI<30
* Able, in the opinion of the investigator, and willing to give informed consent.
* Do not have diagnosed coeliac disease
* Able to understand English

Exclusion Criteria:

Any of the following:

* Urgent, emergency or salvage procedure
* Patients with end stage renal failure defined as an estimated Glomerular Filtration rate (eGFR) <15 mL/min/1.73 m2 calculated from the Modification of Diet in Renal Disease equation,1 or patients who are on long-term haemodialysis or have undergone renal transplantation.
* Patients with persistent or chronic atrial fibrillation.
* Patients with severe liver dysfunction; hepatitis, cirrhosis, jaundice.
* Women who are pregnant or who may become pregnant in the intraoperative period.
* Patients who are participating in another interventional clinical trial.
* Unable, in the opinion of the investigator, or unwilling to give informed consent.
* Have diagnosed coeliac disease
* Unable to understand English

Exclusion criteria for optional MRI research procedure:

* Permanent pacemaker or ICD
* Brain Aneurysm Clip
* Implanted neural stimulator
* Cochlear implant (specific implant must be checked that it is MR safe)
* Ocular foreign body (e.g. metal shavings) unless removed
* Other implanted medical devices: (e.g. Swan Ganz catheter)
* Insulin pump
* Retained metal shrapnel or bullet
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-10-07 (Estimated)

PRIMARY OUTCOMES:
Change of Serum Creatinine level | Baseline, 0-6, 6-12, 24, 48, 72, and up to 96 hours post-operatively
  Measurement of Serum Creatinine level and expressed as umol/L.
Change of Serum Troponin I level | Baseline, 0-6, 6-12, 24, 48 and 72 hours post-operatively
  Measurement of Serum Troponin level and expressed as ng/L.

SECONDARY OUTCOMES:
Post-surgery organ injury: Sepsis-related Organ Failure | Baseline, pre-operatively, 0-6, 6-12, 24, 48, 72 and 96 hours post-operatively
  Sepsis-related Organ Failure Assessment (SOFA) Score. Range 0-3, 3 being the worse score
Post-surgery organ injury: Kidney Injury (Urinary Biomarkers) - NGAL (Neutrophil gelatinase associated lipocalcin) | Baseline, 1 day pre-op, 6-12, 24 and 48 hours post-operatively
  Urine samples will be analysed for biomarkers of renal injury. Measurement of NGAL level will be expressed as μg/L.
Post-surgery organ injury: Kidney Injury (Urinary Biomarkers) - microRNA (Neutrophil gelatinase associated lipocalcin) | Baseline, 1 day pre-op, 6-12, 24 and 48 hours post-operatively
  Urine samples will be analysed for biomarkers of renal injury. Measurement of microRNA in urine samples will be represented by the frequency (%) of identified microRNA.
Post-surgery organ injury: Kidney Injury | Daily for 5 days from Baseline
  Absolute change from baseline for serum creatinine
Post-surgery organ injury: Kidney Injury | At 6 weeks and then 3 months post-surgery
  Serum creatinine and eGFR in all patients using the Modification of Diet in Renal Disease equation. The following is the IDMS-traceable MDRD Study equation (for creatinine methods calibrated to an IDMS reference method) GFR (mL/min/1.73 m2) = 175 × (Scr)-1.154 × (Age)-0.203 × (0.742 if female) × (1.212 if African American) The equation does not require weight or height variables because the results are reported normalized to 1.73 m2 body surface area, which is an accepted average adult surface area.
Post-surgery organ injury: Lung Injury using the Berlin ARDS Score | Baseline, immediately pre-surgery, 0-6, 6-12, 24, 48, 72 and 96 hours post-operatively
  Using the Berlin ARDS score, the measurement of Arterial Alveolar oxygen ratio expressed in kPa/L.
Post-surgery organ injury: GI Tract injury (Biomarker) - AST (Aspartate Transaminase) | Baseline, pre-assessment, pre-operatively, 0-6 and at 6-12, 24, 48, 72 and 96 hours post-operatively.
  Measurement of AST levels in serum and expressed in IU/L. Acute liver injury will be defined as an acute derangement of three times the upper limit of normal.
Post-surgery organ injury: GI Tract injury (Biomarker) - ALT (Alanine Transaminase) | Baseline, pre-assessment, pre-operatively, 0-6 and at 6-12, 24, 48, 72 and 96 hours post-operatively.
  Measurement of ALT levels in serum and expressed in IU/L. Acute liver injury will be defined as an acute derangement of three times the upper limit of normal.
Post-surgery organ injury: GI Tract injury (Biomarker) - Bilirubin | Baseline, pre-assessment, pre-operatively, 0-6 and at 6-12, 24, 48, 72 and 96 hours post-operatively.
  Measurement of Bilirubin levels in serum and expressed in μmol/L. Acute liver injury will be defined as an acute derangement of three times the upper limit of normal.
Post-surgery organ injury: GI Tract injury (Biomarker) - Alkaline Phosphatase | Baseline, pre-assessment, pre-operatively, 0-6 and at 6-12, 24, 48, 72 and 96 hours post-operatively.
  Measurement of Alkaline Phosphatase levels in serum and expressed in IU/L. Acute liver injury will be defined as an acute derangement of three times the upper limit of normal.
Post-surgery organ injury: GI Tract injury (Biomarker) - Serum Amylase | Baseline, pre-assessment, pre-operatively, 0-6 and at 6-12, 24, 48, 72 and 96 hours post-operatively.
  Measurement of Amylase levels in serum and expressed in IU/L. Acute pancreatitis will be defined as a serum amylase concentration >1000 ng/ml.
Assessment of resource use: Extubation | Time (hours) measured from the start of surgery to extubation (up to 30 days)
  Time until extubation
Assessment of resource use: Intensive Care Unit | Time (hours) measured from the start of surgery to discharge from ICU (up to 30 days)
  Length of stay in Intensive Care Unit. Number of hours between admission and discharge from the High Dependency Unit (HDU)
Assessment of resource use: Hospital Stay | Time (days) measured from the start of surgery to discharge from hospital (up to 90 days)
  Length of stay in hospital. Number of days between admission and discharge from the hospital
Clinical events: Sepsis | Time (days) measured from the start of surgery to discharge from hospital (up to 90 days)
  Sepsis will be defined as suspected or documented infection and an acute change in total SOFA score ≥2 points consequent to the infection. For the purposes of the trial suspected or documented infection will be defined as the commencement of intravenous antibiotics. The rise in SOFA score will be assessed within 72 hours of the commencement of antibiotics. Range of SOFA is 0 to 3, 3 being the worse. For the purposes of the study suspected or documented infection will be defined as the commencement of intravenous antibiotics. The rise in SOFA score will be assessed within 72 hours of the commencement of antibiotics.
Clinical events: Peak lactate | Within 24 hours of surgery
  Peak lactate within 24 hours of surgery and time to resolution of hyperlactataemia (arterial serum lactate >2.5 mmol/L) post peak.
Clinical events: Acute Lung Injury | Baseline, immediately pre-surgery, 0-6, 6-12, 24, 48, 72 and 96 hours post-operatively
  Measurement of PaO2/FiO2 ratio and expressed in kPa/L.
Clinical events: Low cardiac output | Time (days) measured from the start of surgery to discharge from hospital (up to 90 days)
  Low cardiac output, defined as new intra-or postoperative intra-aortic balloon pump insertion or a cardiac index of <2.2 L/min/ m2 refractory to appropriate intravascular volume expansion after correction or attempted correction of any dysrhythmias, or the administration of the inotropes Dobutamine, Enoximone, Milrinone or Levosimendan.
Clinical events: Stroke | Time (days) measured from the start of surgery to discharge from hospital (up to 90 days)
  Stroke; diagnosed by brain imaging (CT or MRI), in association with new onset focal or generalized neurological deficit (defined as deficit in motor, sensory or co-ordination functions)
Clinical events: Acute Liver Injury - AST (Aspartate Transaminase) | Time (days) measured from the start of surgery to discharge from hospital (up to 90 days)
  Acute liver injury will be defined as an acute derangement of liver enzymes three times the upper limit of normal, or a serum amylase concentration >1000 ng/m.
Clinical events: Acute Liver Injury - ALT (Alanine Transaminase) | Time (days) measured from the start of surgery to discharge from hospital (up to 90 days)
  Acute liver injury will be defined as an acute derangement of liver enzymes three times the upper limit of normal, or a serum amylase concentration >1000 ng/m.
Clinical events: Acute Liver Injury - Bilirubin | Time (days) measured from the start of surgery to discharge from hospital (up to 90 days)
  Acute liver injury will be defined as an acute derangement of liver enzymes three times the upper limit of normal, or a serum amylase concentration >1000 ng/m.
Clinical events: Acute Liver Injury - Alkaline Phosphatase | Time (days) measured from the start of surgery to discharge from hospital (up to 90 days)
  Acute liver injury will be defined as an acute derangement of liver enzymes three times the upper limit of normal, or a serum amylase concentration >1000 ng/m.
Clinical events: Acute Liver Injury - Serum Amylase | Time (days) measured from the start of surgery to discharge from hospital (up to 90 days)
  Acute liver injury will be defined as an acute derangement of liver enzymes three times the upper limit of normal, or a serum amylase concentration >1000 ng/m.
Clinical events: Acute Intestinal Injury | Time (days) measured from the start of surgery to discharge from hospital (up to 90 days)
  Acute intestinal injury will be defined a radiological, operative or post-mortem evidence of gut ischaemia.
Clinical events: Rate of mortality | Within 30-days from surgery and at 1 year from surgery
  Rate of mortality at 30-days and 1 year from the date of surgery
Clinical events: A composite endpoint Organ Injury, Mortality and Sepsis | Time (days) measured from the start of surgery to discharge from hospital (up to 90 days)
  As above for description of organ injury, mortality and sepsis
Bleeding and Transfusion | Blood loss at 6 hours post-operatively
  The total number of units of red cells and other blood components transfused during the operative period and post-operative hospital stay will be recorded
Mechanism study: Mitochondrial function of microvessels from tissue biopsies | At time of surgery
  50-100 mg biopsies obtained from pedicled left internal mammary artery biopsies. The mitochondrial function will be measured through the Bioenergetic Health Index. The Bioenergetic Health Index (BHI) is calculated using the following formula: BHI=(ATP-linked×reserve capacity)/(proton leak×non-mitochondrial) - as described by Chacko et al. The expected range is 0-100.
Mechanism study: microRNA isolation of microvessels from tissue biopsies | At time of surgery
  The findings will be represented by the frequency (%) of identified microRNA. 50-100 mg biopsies obtained from pedicled left internal mammary artery biopsies.
Mechanism study: Chromatin Immunoprecipitation (ChIP) of microvessels from tissue biopsies | At time of surgery
  To identify protein binding sites that may help identify functional elements in the genome. Findings will be represented by the number (n) of binding sites. 50-100 mg biopsies obtained from pedicled left internal mammary artery biopsies.
Mechanism study: Mitochondrial function measured in right atrium myocardium tissue biopsies | At time of surgery
  50-100 mg myocardial biopsies will be obtained from the right atrium at surgery. The mitochondrial function will be measured through the Bioenergetic Health Index. The Bioenergetic Health Index (BHI) is calculated using the following formula: BHI=(ATP-linked×reserve capacity)/(proton leak×non-mitochondrial) - as described by Chacko et al. The expected range is 0-100.
Mechanism study: microRNA isolation in right atrium myocardium tissue biopsies | At time of surgery
  50-100 mg myocardial biopsies will be obtained from the right atrium at surgery. The findings will be represented by the frequency (%) of identified microRNA.
Mechanism study: Chromatin Immunoprecipitation (ChIP) in right atrium myocardium tissue biopsies | At time of surgery
  50-100 mg myocardial biopsies will be obtained from the right atrium at surgery. To identify protein binding sites that may help identify functional elements in the genome. Findings will be represented by the number (n) of binding sites.
Mechanism study: Mitochondrial function measured in adipose tissue biopsies | At time of surgery
  Adipose tissue collected from epicardial fat at time of surgery. The mitochondrial function will be measured through the Bioenergetic Health Index. The Bioenergetic Health Index (BHI) is calculated using the following formula: BHI=(ATP-linked×reserve capacity)/(proton leak×non-mitochondrial) - as described by Chacko et al. The expected range is 0-100.
Mechanism study: microRNA isolation in adipose tissue biopsies | At time of surgery
  Adipose tissue collected from epicardial fat at time of surgery. The findings will be represented by the frequency (%) of identified microRNA.
Mechanism study: Chromatin Immunoprecipitation (ChIP) in adipose tissue biopsies | At time of surgery
  Adipose tissue collected from epicardial fat at time of surgery. To identify protein binding sites that may help identify functional elements in the genome. Findings will be represented by the number (n) of binding sites.
Mechanism study: Measurement of microvesicles in urine samples | Baseline,1 day before surgery, 6-12, 24 and 48 hours post-operatively.
  Identification of microvesicles. The findings will be represented by the frequency (%) of each identified microvesicle.
Mechanism study: Measurement of microRNA in urine samples | Baseline,1 day before surgery, 6-12, 24 and 48 hours post-operatively.
  The findings will be represented by the frequency (%) of identified microRNA.
Mechanism study: Measurement of histone acetylation in urine samples | Baseline,1 day before surgery, 6-12, 24 and 48 hours post-operatively.
  The findings will be reported as acetylated H3 (ug/mg) over time (hours)
Mechanism study: Measurement of gene expression in urine samples | Baseline,1 day before surgery, 6-12, 24 and 48 hours post-operatively.
  Whole genome sequencing will be achieved through ATAC sequencing. The identified genes will be characterised by average expression count over ATAC.

OTHER OUTCOMES:
Body Composition: Bone Density Scan (DEXA) | Baseline, pre-assessment and 3 months post-surgery
  Assessments of muscle mass/sarcopenia (Appendicular lean mass taken from the DEXA scan)
Imaging Assessment of Cardiometabolic Status: Trans-Oesophageal Echo | At time of surgery
  Diastolic and systolic left ventricular function will be evaluated using intra-operative trans-oesophageal echo in all patients, as per standard care.
Imaging Assessment (optional): Cardiac Magnetic Resonance Imaging - Cardiac Function | Baseline, pre-assessment and 3 months post-surgery
  Assessment of cardiac function, by assessing ventricular function. This will be expressed as ejection fraction (%). Intravenous contrast will be administered via an indwelling venous catheter.
Imaging Assessment (optional): Cardiac Magnetic Resonance Imaging - Cardiac adiposity content | Baseline, pre-assessment and 3 months post-surgery
  Assessment of cardiac adiposity content. A percentage of adipose tissue over total body mass will be calculated. Intravenous contrast will be administered via an indwelling venous catheter.
Imaging Assessment (optional): Cardiac Magnetic Resonance Imaging - Visceral adiposity content | Baseline, pre-assessment and 3 months post-surgery
  Assessment of visceral adiposity content. A percentage of adipose tissue over total body mass will be calculated. Intravenous contrast will be administered via an indwelling venous catheter.
Fitness, Frailty and Muscle Strength: Six Minute Walk Test | Baseline, pre-assessment and 3 months post-surgery
  Fitness will be assessed using the 6-minute walk test (6MWT) which is a standardized test that provides a valid assessment of functional performance. It provides a global assessment of exercise capacity and may better reflect daily activity than more traditional laboratory tests.
Fitness, Frailty and Muscle Strength: Hand Grip Test | Baseline, pre-assessment and 3 months post-surgery
  Hand grip strength will be measured quantitatively by using a dynamometer. The result provides an objective index of general upper body strength and combined with appendicular lean mass (taken from the DEXA scan) could be used to define sarcopenia.
Fitness, Frailty and Muscle Strength: PRISMA-7 Questionnaire | Baseline, pre-assessment and 3 months post-surgery
  Frailty assessment will be by use of the PRISMA-7 Questionnaire. The questions asked are: 1. Are you older than 85 years? 2. Are you male? 3. In general, do you have any health problems that require you to limit your activities? 4. Do you need someone to help you on a regular basis? 5. In general, do you have any health problems that require you to stay at home? 6. If you need help, can you count on someone close to you? 7. Do you regularly use a stick, walker or wheelchair to move about? The participant is asked to answer Yes or No to all 7 questions. SCORING: If the respondent had 3 or more "yes" answers, this indicates an increased risk of frailty and the need for further clinical review.
Activity Levels and Sleep: Accelerometer Assessments | Baseline, pre-assessment and 3 months post-surgery
  Activity levels and sleep are measured by the use of seven day accelerometer assessments
Comorbidity and Inflammation - CRP (C-Reactive-Protein) assay (Abcam) | Baseline, pre-assessment and 3 months post-surgery
  Pre-existing inflammation, renal impairment and heart failure will be assessed using highly sensitive CRP assay, NT-proBNP (both Abcam), and estimated Glomerular Filtration Rate (from serum creatinine). The acceptable range for CRP values using the abcam kit is 34.29 - 25,000 pg/mL. For values above 25ng/mL, the samples will be diluted and re-assayed. Samples < 34.29 pg/mL will be re-assayed at higher concentration when possible; otherwise the concentrations will be accepted if higher than assay detection limit (2 pg/L). For samples <2pg/mL a no-expression value will be assigned.
Comorbidity and Inflammation - NT-proBNP (Abcam) | Baseline, pre-assessment and 3 months post-surgery
  Pre-existing inflammation, renal impairment and heart failure will be assessed using highly sensitive CRP assay, NT-proBNP (both Abcam), and estimated Glomerular Filtration Rate (from serum creatinine). The acceptable range for NT-proBNP values using the abcam kit is 0.14 - 100 ng/mL. For values above 100ng/mL, the samples will be diluted and re-assayed. Samples < 0.14 ng/mL will be re-assayed at higher concentration when possible; otherwise a no-expression value will be assigned.
Comorbidity and Inflammation - estimated Glomerular Filtration Rate | Baseline, pre-assessment and 3 months post-surgery
  Pre-existing inflammation, renal impairment and heart failure will be assessed using highly sensitive CRP assay, NT-proBNP (both Abcam), and estimated Glomerular Filtration Rate (from serum creatinine). Formula for GFR (mL/min/1.73 m2) = 175 × (Scr)-1.154 × (Age)-0.203 × (0.742 if female) × (1.212 if African American) The equation does not require weight or height variables because the results are reported normalized to 1.73 m2 body surface area, which is an accepted average adult surface area.
Endothelial function: Blood samples | Baseline, 6-12 and 48 hours post-surgery
  Markers of endothelial activation will be measured in blood samples using flow cytometry.
Endothelial function: Reactive Hyperaemia Peripheral Arterial Tonometry (RH-PAT) | 1 day before surgery and 24 hours post-surgery
  Regional endothelial dysfunction will be measured as the reactive hyperaemia peripheral arterial tonometry (RH-PAT) index using the Endo-PAT 2000 (Itamar Medical Ltd., Caesarea, Israel)
Endothelial function: Global endothelial dysfunction | End of surgery, 0-6, 6-12, 24, 48, 72 and 96 hours post-operatively (until the timepoint serum arterial lactate falls below 2.5 mmol/L)
  Global endothelial dysfunction will also be measured indirectly as the measured time to resolution of oxygen debt defined as the period of time from the end of surgery until the measured serum arterial lactate level falls below 2.5 mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin J Murphy, MD, Study Chair — BHF Professor of Cardiac Surgery, University of Leicester; Mustafa Zakkar, PhD, Principal Investigator — Associate Professor, University of Leicester
Locations (1):
- University of Leicester, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No